CLINICAL TRIAL: NCT01754012
Title: New Dietary Strategies Addressing the Specific Needs of Elderly Population for an Healthy Aging in Europe
Brief Title: European Project on Nutrition in Elderly People
Acronym: NU-AGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Claudio Franceschi, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 266486
Record Dates: First submitted 2012-12-09; First posted 2012-12-21 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Aging
Keywords: Nutrition; Dietary intervention; Aging; Inflammation; Elderly; Europe
MeSH Terms: conditions — Inflammation | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Intervention (Experimental): This group will follow for a year the NU-AGE whole diet approach elderly-specific and will be supplemented with 10micrograms per day of Vitamin D (cholecalciferol) from MCOHealth.
  Interventions: Dietary Supplement: Dietary Intervention
- Control Group (No Intervention): This group will follow the habitual diet.

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — nutrient-rich diet and 10micrograms per day of Vitamin D (cholecalciferol) supplement from MCOHealth
  Other Names: NU-AGE diet; NU-AGE whole diet approach
  Arms: Dietary Intervention

SUMMARY:
NU-AGE is a large multidisciplinary consortium (31 partners, from 17 EU countries) involving nutritionists, bio-gerontologists, immunologists and molecular biologists from the most prestigious institutions in Europe, 5 large food industries, 8 traditional food companies and 1 biotech SME, SPES GEIE and CIAA, covering the SME Food Industrial Associations of 13 European countries and the European Confederation the food and drink industry. NU-AGE aims are: 1. to counteract the physical/cognitive decline occurring in the elderly as a consequence of the progressive alteration of different organs/systems (immune and cardiovascular systems, bone, brain, muscle and intestine) by one year elderly-tailored whole diet intervention on 1250 healthy elderly men and women aged 65-79 years (half diet, half control) from 5 different EU regions; 2. to assess the effect of the newly designed food pyramid specific for 65+ EU citizens on the different organs/systems using a large set of biomarkers related to nutrition and aging, with particular attention to the low grade, chronic, systemic inflammatory status named inflammageing, a major risk factor for common age-related diseases; 3. to perform in a subgroup of 120 subjects in depth studies and high throughput "omics" to identify cellular/molecular targets/mechanisms responsible for whole diet effect; 4. to perform genetic and epigenetic studies to assess the role of individual variability on the response to diet; 5. to adopt an integrative comprehensive approach (systems biology) to analyze the whole set of data. The results of dietary intervention will be used to develop elderly-tailored prototypes of functional foods and to improve traditional foods. The research activity will be accompanied and followed by a strong activity of dissemination and industrial exploitation to support EU strategies on nutritional recommendations, thus contributing to the implementation of legislation related to nutritional and health claims for elderly in Europe.

ELIGIBILITY:
Inclusion Criteria:

* 65-79 years old.
* Free of clinically diagnosed overt disease for at least 2 years.
* Free-living, independent.

Exclusion Criteria:

* <65 or > 79 years old.
* Overt disease such as aggressive cancer or dementia.
* Unstable organ failure or organ failure necessitating a special diet.
* Heart failure.
* Renal failure.
* Respiratory failure.
* Liver failure.
* Type 1 diabetes mellitus.
* Chronic use of corticosteroids.
* Recent (previous 2 months) use of antibiotics.
* Recent (previous 3 months) change to habitual medication (e.g statins and thyroxine) use
* Presence of food allergy/intolerance or disease necessitating a special diet.
* Malnutrition, as diagnosed by body mass index < 18.5 kg/m2.
* Body weight loss of >10% BW within 6 months.
* Presence of frailty (as assessed by the presence of at least three out of five criteria according to Fried et al., 2001: unintentional weight loss, self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity).
* Individual unable to give informed consent.
* Volunteers showing previously unrecognized illness will also be excluded.

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Inflammatory Response | 1 year
  Reduction of inflammatory markers after one-year of NU-AGE dietary intervention in elderly.
  Measures of inflammatory status and immune health will be evaluated on plasma: C-reactive protein (hsCRP) IL-1Beta, IL-12, INF gamma, IL-6, sIL-6R, IL-1RA, TNFalpha, IL-17, IL-8, IL-10, TGF-beta1, positivity for HCMV.

SECONDARY OUTCOMES:
Cognitive Status | 1 year
  The following standardized questionnaires will be administered to volunteers pre and post dietary intervention to evaluate cognitive function:
  1. CERAD Neuropsychological Assessment Battery
  2. Domain Specific Tests (GDS, Babcock story Recall, Trail Making Test)
Cardiovascular Health Status | 1 year
  Evaluation of blood pressure and measure of lipid profile (triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol) pre and post dietary intervention on plasma.
Insulin sensitivity | 1 year
  Glucose, insulin and Hba1C will be measured on plasma pre and post dietary intervention
Liver Function Status | 1 year
  ASAT, ALAT, GGT and alkaline phosphatase parameters will be measured on plasma samples pre and post dietary intervention.
Hormonal Status | 1 year
  Leptin and adiponectin hormones will be measured on plasma samples pre and post dietary intervention
Nutritional Status | 1 year
  The Nutritional status will be evaluated on plasma measuring vitamin B12 and folate concentrations.
Digestive Health Status | 1 year
  Questionnaire to assess bowel function, gastrointestinal disturbances and evacuation frequency will be administered to participants pre and post dietary intervention.
Bone Health Status | 1 year
  All participants, pre and post dietary intervention, will undergone DXA exam to evaluate bone mineral density, also 25-OH vitamin D, parathyroid hormone will be measured on plasma samples.
Physical Functioning | 1 year
  The following standardized questionnaires will be administered to volunteers pre and post dietary intervention to evaluate physical function:
  1. SPPB
  2. Hand grip test
  3. Gait Speed Test
  4. ADL, IADL
  5. PASE
Changes on Cellular and Molecular mechanisms after diet: Immunological Status | 1 year
  On a subgroup of 125subjects (pre and post diet), the following of additional analyses on plasma will be performed to evaluate the immunological status of participants:
  1. Expression and responsiveness of Toll-like receptors, measured as production of downstream cytokines (IFN-a, IFN-b, IFN-y, IL12p40, IL12p70, SOCS3)
  2. Expression of co-stimulatory molecules (CD1, MHC Class II, CD40, CD80, CD86, CD152, CD154, DC1/DC2)
Changes on Cellular and Molecular mechanisms after diet: Epigenetic signature | 1 year
  On a subgroup of 120 subjects (pre and post diet), the epigenetic signature will be evaluated through methylation assay on isolated PBMC.
Changes on Cellular and Molecular mechanisms after diet: biochemical modifications | 1 year
  On a subgroup of 120 subjects (pre and post diet), proteasome and immunoproteasome composition and activity will be measured on proteins from isolated PBMC.
Transcriptomics | 1 year
  On a subgroup of 120 subjects (pre and post diet) a transcriptomics analysis will be performed on mRNA from isolated PBMC by high throughput technologies "omics".
Metabolomics | 1 year
  On a subgroup of 120 subjects (pre and post diet) a the metabolic profile will be performed on urine and plasma/serum by high throughput technologies "omics".
Metagenomics | 1 year
  On a subgroup of 120 subjects (pre and post diet) the functional and compositional analysis of the microbiota will be assessed on feces by high throughput technologies "omics".

OTHER OUTCOMES:
Habitual Diet | 4 months
  Over the course of the 1-year intervention period assessment of habitual diet, will be conducted by repeated the 7 days nutritional diary administered in person (month 1 and 12) and 3 days nutritional diary administered at interim time points (months 4-8) by telephone.
Genetic profiling | Time 0
  The genetic profiling of genes involved in inflammageing will be analyzed (only before diet) in order to assess genotype-phenotype and genotype-diet phenotype associations.
General Health information | 1 year
  Information will be collected at month 1 and 12 on smoking status, health status, physical activity levels, alcohol consumption and medication and supplement use, so that these parameters can be added to all statistical analysis models as confounders

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Franceschi, MD, Principal Investigator — University of Bologna
Locations (5):
- Auvergne Research Center on Human Nutrition, Clermont-Ferrand, France
- University of Bologna-Department of Speciality, Diagnostic and Experimental Medicine, Bologna, Bologna, Italy
- University of Wageningen-Division of Human Nutrition, Wageningen, Netherlands
- Warsaw University of Life Science SGGW-WULS-Department of Human Nutrition, Warsaw, Poland
- Department of Nurition-University of East Anglia, Norwich, United Kingdom

REFERENCES:
- [Derived] Grootswagers P, Mensink M, Berendsen AAM, Deen CPJ, Kema IP, Bakker SJL, Santoro A, Franceschi C, Meunier N, Malpuech-Brugere C, Bialecka-Debek A, Rolf K, Fairweather-Tait S, Jennings A, Feskens EJM, de Groot LCPGM. Vitamin B-6 intake is related to physical performance in European older adults: results of the New Dietary Strategies Addressing the Specific Needs of the Elderly Population for Healthy Aging in Europe (NU-AGE) study. Am J Clin Nutr. 2021 Apr 6;113(4):781-789. doi: 10.1093/ajcn/nqaa368. PMID 33515034
- [Derived] Jennings A, Tang J, Gillings R, Perfecto A, Dutton J, Speakman J, Fraser WD, Nicoletti C, Berendsen AAM, de Groot LCPGM, Pietruszka B, Jeruszka-Bielak M, Caumon E, Caille A, Ostan R, Franceschi C, Santoro A, Fairweather-Tait SJ. Changing from a Western to a Mediterranean-style diet does not affect iron or selenium status: results of the New Dietary Strategies Addressing the Specific Needs of the Elderly Population for Healthy Aging in Europe (NU-AGE) 1-year randomized clinical trial in elderly Europeans. Am J Clin Nutr. 2020 Jan 1;111(1):98-109. doi: 10.1093/ajcn/nqz243. PMID 31559434
- [Derived] Giampieri E, Ostan R, Guidarelli G, Salvioli S, Berendsen AAM, Brzozowska A, Pietruszka B, Jennings A, Meunier N, Caumon E, Fairweather-Tait S, Sicinska E, Feskens EJM, de Groot LCPGM, Franceschi C, Santoro A. A Novel Approach to Improve the Estimation of a Diet Adherence Considering Seasonality and Short Term Variability - The NU-AGE Mediterranean Diet Experience. Front Physiol. 2019 Mar 5;10:149. doi: 10.3389/fphys.2019.00149. eCollection 2019. PMID 30890946
- [Derived] Pujos-Guillot E, Petera M, Jacquemin J, Centeno D, Lyan B, Montoliu I, Madej D, Pietruszka B, Fabbri C, Santoro A, Brzozowska A, Franceschi C, Comte B. Identification of Pre-frailty Sub-Phenotypes in Elderly Using Metabolomics. Front Physiol. 2019 Jan 24;9:1903. doi: 10.3389/fphys.2018.01903. eCollection 2018. PMID 30733683
- [Derived] Jennings A, Berendsen AM, de Groot LCPGM, Feskens EJM, Brzozowska A, Sicinska E, Pietruszka B, Meunier N, Caumon E, Malpuech-Brugere C, Santoro A, Ostan R, Franceschi C, Gillings R, O' Neill CM, Fairweather-Tait SJ, Minihane AM, Cassidy A. Mediterranean-Style Diet Improves Systolic Blood Pressure and Arterial Stiffness in Older Adults. Hypertension. 2019 Mar;73(3):578-586. doi: 10.1161/HYPERTENSIONAHA.118.12259. PMID 30636547
- [Derived] Ostan R, Guidarelli G, Giampieri E, Lanzarini C, Berendsen AAM, Januszko O, Jennings A, Lyon N, Caumon E, Gillings R, Sicinska E, Meunier N, Feskens EJM, Pietruszka B, de Groot LCPGM, Fairweather-Tait S, Capri M, Franceschi C, Santoro A. Cross-Sectional Analysis of the Correlation Between Daily Nutrient Intake Assessed by 7-Day Food Records and Biomarkers of Dietary Intake Among Participants of the NU-AGE Study. Front Physiol. 2018 Oct 1;9:1359. doi: 10.3389/fphys.2018.01359. eCollection 2018. PMID 30327612
- [Derived] Maijo M, Ivory K, Clements SJ, Dainty JR, Jennings A, Gillings R, Fairweather-Tait S, Gulisano M, Santoro A, Franceschi C, Carding SR, Nicoletti C. One-Year Consumption of a Mediterranean-Like Dietary Pattern With Vitamin D3 Supplements Induced Small Scale but Extensive Changes of Immune Cell Phenotype, Co-receptor Expression and Innate Immune Responses in Healthy Elderly Subjects: Results From the United Kingdom Arm of the NU-AGE Trial. Front Physiol. 2018 Jul 26;9:997. doi: 10.3389/fphys.2018.00997. eCollection 2018. PMID 30093866
- [Derived] Jennings A, Cashman KD, Gillings R, Cassidy A, Tang J, Fraser W, Dowling KG, Hull GLJ, Berendsen AAM, de Groot LCPGM, Pietruszka B, Wierzbicka E, Ostan R, Bazzocchi A, Battista G, Caumon E, Meunier N, Malpuech-Brugere C, Franceschi C, Santoro A, Fairweather-Tait SJ. A Mediterranean-like dietary pattern with vitamin D3 (10 microg/d) supplements reduced the rate of bone loss in older Europeans with osteoporosis at baseline: results of a 1-y randomized controlled trial. Am J Clin Nutr. 2018 Sep 1;108(3):633-640. doi: 10.1093/ajcn/nqy122. PMID 30007343
- [Derived] Marseglia A, Xu W, Fratiglioni L, Fabbri C, Berendsen AAM, Bialecka-Debek A, Jennings A, Gillings R, Meunier N, Caumon E, Fairweather-Tait S, Pietruszka B, De Groot LCPGM, Santoro A, Franceschi C. Effect of the NU-AGE Diet on Cognitive Functioning in Older Adults: A Randomized Controlled Trial. Front Physiol. 2018 Apr 4;9:349. doi: 10.3389/fphys.2018.00349. eCollection 2018. PMID 29670545
- [Derived] Fairweather-Tait SJ, Jennings A, Harvey LJ, Berry R, Walton J, Dainty JR. Modeling tool for calculating dietary iron bioavailability in iron-sufficient adults. Am J Clin Nutr. 2017 Jun;105(6):1408-1414. doi: 10.3945/ajcn.116.147389. Epub 2017 Apr 5. PMID 28381473
- [Derived] Hooper L, Bunn DK, Abdelhamid A, Gillings R, Jennings A, Maas K, Millar S, Twomlow E, Hunter PR, Shepstone L, Potter JF, Fairweather-Tait SJ. Water-loss (intracellular) dehydration assessed using urinary tests: how well do they work? Diagnostic accuracy in older people. Am J Clin Nutr. 2016 Jul;104(1):121-31. doi: 10.3945/ajcn.115.119925. Epub 2016 May 25. PMID 27225436
- [Derived] Hooper L, Abdelhamid A, Ali A, Bunn DK, Jennings A, John WG, Kerry S, Lindner G, Pfortmueller CA, Sjostrand F, Walsh NP, Fairweather-Tait SJ, Potter JF, Hunter PR, Shepstone L. Diagnostic accuracy of calculated serum osmolarity to predict dehydration in older people: adding value to pathology laboratory reports. BMJ Open. 2015 Oct 21;5(10):e008846. doi: 10.1136/bmjopen-2015-008846. PMID 26490100
- [Derived] Berendsen A, Santoro A, Pini E, Cevenini E, Ostan R, Pietruszka B, Rolf K, Cano N, Caille A, Lyon-Belgy N, Fairweather-Tait S, Feskens E, Franceschi C, de Groot CP. Reprint of: A parallel randomized trial on the effect of a healthful diet on inflammageing and its consequences in European elderly people: design of the NU-AGE dietary intervention study. Mech Ageing Dev. 2014 Mar-Apr;136-137:14-21. doi: 10.1016/j.mad.2014.03.001. Epub 2014 Mar 20. PMID 24657127
- [Derived] Hooper L, Bunn D, Jimoh FO, Fairweather-Tait SJ. Water-loss dehydration and aging. Mech Ageing Dev. 2014 Mar-Apr;136-137:50-8. doi: 10.1016/j.mad.2013.11.009. Epub 2013 Dec 9. PMID 24333321
- [Derived] Fairweather-Tait SJ, Wawer AA, Gillings R, Jennings A, Myint PK. Iron status in the elderly. Mech Ageing Dev. 2014 Mar-Apr;136-137:22-8. doi: 10.1016/j.mad.2013.11.005. Epub 2013 Nov 22. PMID 24275120